CLINICAL TRIAL: NCT02705612
Title: Efficacy and Safety of Radiotherapy Concurrently Combined With Cisplatin and Nimotuzumab for Patients With Locally Advanced Cervical Cancer
Brief Title: Phase II Clinical Trial of Concurrent Chemoradiotherapy Combined Nimotuzumab for Stage IIB-IVA Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Mei Shi, Director and professor of Radiation Oncology，Xijing Hospital，Fourth Millitary Medical University, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJFL-2016-02-LACC-Nimotuzumab
Record Dates: First submitted 2016-03-05; First posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer; cisplatin; nimotuzumab
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Brachytherapy; nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (Other): Patients receive cisplatin IV over 60-90 minutes on days 1, 8, 15, 22, and 29. Patients also undergo external-beam radiation therapy once daily, 5 days a week, for approximately 5 weeks. Patients then undergo high-dose rate intracavitary brachytherapy.
  Interventions: Drug: Cisplatin; Radiation: External Beam Radiation Therapy; Radiation: Internal Radiation Therapy
- experimental group (Experimental): Patients receive cisplatin and undergo external-beam radiation and brachytherapy as the patients in control group. Patients also receive nimotuzumab during the external radiotherapy.
  Interventions: Drug: Cisplatin; Radiation: External Beam Radiation Therapy; Radiation: Internal Radiation Therapy; Drug: nimotuzumab

INTERVENTIONS:
Drug: Cisplatin
Radiation: External Beam Radiation Therapy
Radiation: Internal Radiation Therapy
Drug: nimotuzumab
  Arms: experimental group

SUMMARY:
The purpose of this phase II trial is to determine the feasibility and efficacy of nimotuzumab injection combined with concurrent chemoradiotherapy for initially inoperable locally advanced cervical cancer.

DETAILED DESCRIPTION:
For locally advanced cervical cancer, radical radiation with concurrent chemotherapy remains the standard treatment recommended by NCCN. However, in more than 35% of cases, tumor persistence recurrence or metastasis would occur after chemoradiation. Nimotuzumab, belongs to anti-EGFR monoclonal antibodies, has proved to be useful in multiple solid tumors, such as NPC, colorectal cancer, etc.

In recent years, nimotuzumab was also applied in recurrence or metastasis cervical cancer. It was proved to be well tolerated and might have a role in the treatment of advanced cervical cancer. However, there is no publication about nimotuzumab used in locally advanced cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years to 70 Years，female
* Histological diagnosis of squamous cell carcinoma of cervix, FIGO stage IIB-IVA,with diameter 4-6 cm, without distant metastasis.
* no chance of surgery confirmed by more than two deputy chief doctors of gynecology.
* Moderate or high expression of EGFR
* The function of main organ is normal, including blood, heart, lung, liver, and kidney. Without history of hypertension, stroke. Blood pressure is normal before treatment.
* WBC≥3.5×10E9/L，ANC≥1.5×10E9/L；HB≥90g/L，PLT≥100×10E9/L
* ALT, AST and Cr below 1.5 times of normal level
* Willing to accept treatment
* Ability to comply with trial requirements KPS≥70

Exclusion Criteria:

* Evidence of distance metastasis
* Impossible to measure the diameter of tumor, or the tumor is too huge (diameter>6cm)
* Couldn't examine with pelvic MRI due to a variety of reasons
* Used to treat with radiotherapy chemotherapy or molecular target therapy and immune therapy
* Diagnosed with another malignant tumor in 5 years
* Used to be a volunteer of other clinical trial.
* Used to be allergic reaction with grade 3 or 4 degree to any experimental drugs
* Severe medical history of lung ,liver, kidney or heart.
* Active infection in any part of the whole body.
* Examination results showed radiotherapy contraindications

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | at 3 years
  Described with Kaplan-Meier curves and unadjusted logrank tests.
disease free survival rate | at 3 years
non-distant metastasis survival rate | at 3 years
survival period of non-progressive. | at 3 years

SECONDARY OUTCOMES:
Quality of life | 3 years
Radiation protocol compliance | 3 years
Rate of acute and long-term toxicities | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mei Shi, MD, Principal Investigator — department of radiation oncology
Locations (1):
- Department of Radiation Oncology, Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China